CLINICAL TRIAL: NCT06765005
Title: A Phase Ib/II.a Clinical Study of the Safety, Pharmacokinetics and Preliminary Efficacy of MG-K10Humanized Monoclonal Antibody Injection in Adolescent Patients with Moderate to Severe Atopic Dermatitis Aged 12-18 Years.
Brief Title: IB/IIa Study of MG-K10 in Adolescent Moderately Severe Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-K10-AD-004
Record Dates: First submitted 2024-07-12; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Drug dosage: 600mg for the first time, 300mg for the next time, subcutaneous injection, divided into 2 groups, every 2 weeks for a total of 4 doses, every 4 weeks for a total of 2 doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MG-K10 Regimen 1 (Experimental): Subcutaneous injection, once every 2 weeks
  Interventions: Drug: MG-K10

INTERVENTIONS:
Drug: MG-K10 — Subcutaneous injection, once every 4 weeks

SUMMARY:
This study was designed to reflect the safety pharmacokinetics and preliminary efficacy of MG-K10 Humanized Monoclonal Antibody Injection in adolescent patients 12-18 weeks of age with moderate to severe atopic dermatitis, administered every 2 or 4 weeks for 8 weeks

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the MG-K10 humanized monoclonal antibody injection in adolescent moderate-to-severe atopic dermatitis (AD) patients.

Secondary Objective:

To evaluate the pharmacokinetic (PK) profile, preliminary efficacy, and safety of MG-K10 humanized monoclonal antibody injection in adolescent patients with moderate-to-severe AD.To assess the pharmacokinetic (PK) profile, preliminary efficacy, pharmacokinetic (PD) profileand immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years old ≤ <18 years old (based on the date of signing the ICF), regardless of gender.

   Body weight ≥ 30 kg;
2. patients with a diagnosis of AD that meets the American Academy of Dermatology Consensus Criteria (2014), with a diagnosis of AD or history of eczema ≥6 months prior to screening, and with the following criteria

2. Patients with a diagnosis of AD that meets the American Academy of Dermatology Consensus Criteria (2014), a history of AD or eczema ≥ 6 months prior to screening, and the following criteria:

* EASI ≥16 at screening and baseline;
* EASI ≥16 at Screening and Baseline; IGA ≥3 at Screening and Baseline;
* BSA involvement in skin lesions ≥10% at Screening and Baseline; 3. determined within 6 months prior to Screening to be inadequately treated with topical medications or medically inappropriate for treatment with topical medications; andmedically inappropriate for treatment with topical medications (e.g., significant side effects or safety risks).

  (e.g., significant side effects or safety risks);

Inadequate efficacy is defined as:

- At least 4 weeks of potent or 2 weeks of ultra-potent topical glucocorticosteroids or 4 weeks of topical calcitonin within 6 months prior to Screening.Inadequate treatment outcome is defined as or maintain a state of remission or low disease activity (equivalent to an IGA score of 0 [=(equivalent to an IGA score of 0 [= asymptomatic] - 2 [= mildly symptomatic]);- Important side effects or safety risks are those that, as assessed by the investigator or the patient's treating physician, outweigh the potential therapeutic benefit.Important side effects or safety risks are those that, as assessed by the investigator or the patient's treating physician, outweigh the potential therapeutic benefit, including treatment intolerance Important side effect or safety risk means a side effect or risk that outweighs the potential therapeutic benefit, as assessed by the Investigator or the patient's treating physician, including treatment intolerance, allergic reaction, significant skin atrophy, and systemic reaction。 4. Subjects of potential reproductive potential (e.g., women who have had their first menstruation or men who have had spermatozoa) must agree to and comply with the use of effective contraception throughout the study period and for 6 months after the last dose.Subjects of potential reproductive potential (e.g., women who have had their first period or men who have had spermatozoa) must agree to and comply with effective contraception throughout the study period and for 6 months after the last dose.

5. the subject and/or the subject's parent or other legal guardian voluntarily signs a written informed consent form and is able to communicate with the investigator.

Subjects and/or their parents or other legal guardians voluntarily sign a written informed consent form and are able to communicate well with the investigator and comply with protocol requirements for follow-up visits.

Exclusion Criteria:

1. Individuals with severe allergic reactions to the test drug or its analogs; those who cannot administer subcutaneous injections, e.g., those on anticoagulant therapy, known bleeding disorders, or idiopathic thrombocytopenic purpura;
2. Presence of other active skin conditions (e.g., psoriasis or lupus erythematosus) that may affect AD evaluation;
3. Presence of diseases that may require systemic hormonal or immunosuppressive therapy;
4. Patients with ocular disease that, in the judgment of the investigator, is not appropriate for enrollment, such as a previous history of atopic keratoconjunctivitis with involvement of the cornea; an ophthalmologist will be required to make a diagnosis if the investigator is unable to make a determination;
5. Use of targeted inhibitors (e.g., JAK inhibitors), systemic glucocorticoids, cyclosporine, or other immunosuppressants (e.g., methotrexate) within 4 weeks prior to randomization systemic glucocorticoids, cyclosporine or other immunosuppressive agents (e.g., methotrexate, mycophenolate mofetil, azathioprine, etc.), phosphodiesterase (PDE4) inhibitors, ultraviolet (UV) radiation, and other immunosuppressive agents.

   Systemic glucocorticoids, cyclosporine or other immunosuppressants (e.g., methotrexate, mycophenolate mofetil, and azathioprine), phosphodiesterase (PDE4) inhibitors, ultraviolet radiation therapy, systemic AD Cyclosporine or other immunosuppressants (methotrexate, mycophenolate mofetil, and azathioprine), phospholipase (PDE4) inhibitors, ultraviolet radiation therapy, and systemic herbal medicine for AD Have used a biologic within 10 weeks prior to randomization or have not exceeded 5 half-lives (whichever is longer).

   have used a biologic agent within 10 weeks prior to randomization or have not exceeded 5 half-lives, whichever is longer;)

   -Allergen-specific immunotherapy in the 6 months prior to randomization;
6. Those who stopped all topical medications for less than 2 weeks prior to randomization, including topical glucocorticoids, topical calcium-modulated phosphatase inhibitors, antibiotic-complexed creams, and topical herbal treatments;
7. Participated in a clinical study with a biologic within 3 months or 5 half-lives, whichever is longer, prior to screening; participated in a clinical study with a biologic within 1 month or 5 half-lives, whichever is longer, prior to randomization.

   Participated in a clinical study with a biologic agent within 3 months or 5 half-lives, whichever is longer, prior to screening; participated in a clinical study with a non-biologic agent within 1 month or 5 half-lives, whichever is longer, prior to randomization.

   Participated in a clinical study of a non-biologic agent drug within 1 month or 5 half-lives, whichever is longer, prior to randomization, or plans to participate in a clinical study of another drug during the study period.

   Participated in a clinical study of a non-biologic agent drug within 1 month or 5 half-lives, whichever is longer, prior to randomization, or plan to participate in a clinical study of another drug during the study period.

   Subjects who have participated in a clinical study of this product; subjects who have used monoclonal antibodies to the interleukin 4 receptor alpha subunit (IL-4Rα) and, in the judgment of the investigator, have developed resistance or serious drug-related AEs.

   Subjects who, in the judgment of the Investigator, have developed drug resistance or severe drug-related AEs;
8. Those who have received live/live attenuated vaccine within 3 months prior to screening or plan to do so during the study;
9. Persons with chronic active infections or acute infections requiring systemic (oral and intravenous) antipathogenic microbial (anti-bacterial, viral, fungal, etc.) therapy within 4 weeks prior to randomization;
10. Evidence of active tuberculosis or previous evidence of active tuberculosis without appropriate documented treatment; active tuberculosis infection as indicated by chest X-ray (frontal and lateral) or CT, etc., within 3 months prior to/screening period;
11. History of parasitic infection within 6 months prior to screening;
12. Patients with a history of malignant tumors;
13. Comorbidities of other serious diseases, including but not limited to cardiovascular, metabolic, and neurological diseases, which are assessed by the investigator to be unsuitable for immunosuppressive therapy;
14. Those who, in the opinion of the investigator, have other conditions that make them unsuitable for participation in the study;
15. History of alcohol or drug abuse within 6 months prior to screening;

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | up to 113 days
  security

SECONDARY OUTCOMES:
PK finish line | up to 113 days
  PK endpoint: MG-K10 blood concentration
PK finish line | up to 147 days
  Cmax
PK finish line | 21week
  AUC
Percentage of subjects with an overall investigator-assessed IGA score | 8 weeks after administration
  Percentage of subjects with an overall investigator-assessed IGA score of 0 or 1 from baseline at each evaluation visit site;
Percentage of subjects with an overall investigator-assessed IGA score decrease of ≥2 points from baseline at each evaluation visit site; | 8 weeks after administration
  Effectiveness
The changes in eczema area at each evaluation visit point compared with the baseline. | up to 113 days
  Change from baseline and rate of change in eczema area and severity index (EASI) score at each evaluation visit site;
Percentage of subjects achieving EASI-50, EASI-75, and EASI-90 at each evaluation visit site; | up to 113 days
  Percentage of subjects achieving EASI-50, EASI-75, and EASI-90 (≥ 50% / 75% / 90% reduction in EASI score from baseline) at each evaluation visit viewpoint;
Change from baseline in weekly mean NRS | up to 113 days
  Change from baseline and rate of change in weekly mean of daily peak itch score（Numerical rating scale 0-10）;
Change from baseline in weekly mean NRS score | up to 113 day
  Percentage of subjects whose weekly mean daily peak itch score （Numerical rating scale 0-10）decreased by ≥4 points from baseline;
Change in BSA from baseline | up to 113 days
  Change from baseline and rate of change in body surface area (BSA) involved in skin lesions at each evaluation visit site;
(POEM) score change from baseline | up to 113 days
  Change from baseline in patient eczema self-assessment (POEM) scores at each evaluation visit site;

CONTACTS AND LOCATIONS:
Overall Officials: liming wu, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital;, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We may work with other companies to develop follow-up clinical programs in China or global clinical programs